CLINICAL TRIAL: NCT06883981
Title: Capturing Autobiographical Memory Formation in People Moving Through Real-World Spaces Using Synchronized Wearables and Intracranial Recordings of EEG
Brief Title: Capturing Autobiographical Memory Formation in Real World Spaces Using Multimodal Recordings
Acronym: CAPTURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH); University of California, San Diego (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Cory Inman, Assistant Professor, University of Utah
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00183967; 1R61MH135109-01 (NIH)
Record Dates: First submitted 2025-03-10; First posted 2025-03-19 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy; Autobiographical Memory
Keywords: Autobiographical memory; Memory; IEEG; Epilepsy; Real-World Navigation; Spatial Memory; Hippocampus; Medial Temporal Cortex; Multi-Modal Recording
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuroethical Assessment Group (No Intervention): Patients with epilepsy who have Neuropace RNS implants who will be surveyed about the neuroethics of real-world multi-modal recordings to assess their attitude toward research data sharing and confidentiality.
- Multi-Modal Recording System Assessment Group (Experimental): Patients with epilepsy who have Neuropace RNS implants, and patients without epilepsy/RNS implants, who will participate in real-world navigation and autobiographical memory tasks in order to evaluate the reliability and signal quality of the multi-modal recording system.
  Interventions: Behavioral: Free and Cued Recall Memory. Temporal Sequence and Spatial Memory

INTERVENTIONS:
Behavioral: Free and Cued Recall Memory. Temporal Sequence and Spatial Memory — Memory for real-world episodic experiences will be tested in the laboratory first with free recall (spoken narration of their recollections from each environment) and then with cued recall, in which participants will be cued with an event image from the CAPTURE app, a map location, or a relative time and asked to recall the other two non-cued pieces of episodic information (event, place, or time). Because we will know the 'ground truth', the cued recall test will allow us to measure how accurately the participant is able to remember key details of each episode. We will also assess temporal order memory by asking participants to arrange 1st person images in the order in which they occurred, and we will assess spatial memory by asking them to place each image on a schematic map of the venue.
  Arms: Multi-Modal Recording System Assessment Group

SUMMARY:
The goal of this observational study is to develop novel methods for integrating multimodal data streams with invasive neural recordings to study autobiographical memory (AM) formation in individuals with implanted neurostimulation devices (e.g., NeuroPace RNS) for epilepsy treatment. The main questions it aims to answer are:

How does the brain encode and retrieve real-world autobiographical memories? Can multimodal data integration enhance our understanding of memory-related cognitive and neural mechanisms?

Participants will:

* Use a smartphone-based recording application (CAPTURE app) to collect real-world data.
* Have their wearable sensor data (e.g., audio-visual, accelerometry, GPS, autonomic physiology, eye tracking) synchronized with invasive neural recordings.

Researchers will analyze these multimodal data streams to develop new analytic approaches for studying memory formation in naturalistic settings, with the long-term goal of informing neuromodulation-based memory enhancement treatments for individuals with memory disorders.

DETAILED DESCRIPTION:
This observational study aims to develop and validate novel methodologies for integrating multimodal data streams with invasive neural recordings in individuals with implanted neurostimulation devices (e.g., NeuroPace RNS) undergoing treatment for epilepsy. The study focuses on understanding the neural mechanisms underlying autobiographical memory (AM) formation and retrieval in real-world settings. By leveraging real-time, ecologically valid data collection, this research seeks to bridge the gap between controlled laboratory-based memory studies and naturalistic memory processes.

Study Design and Data Collection Participants with implanted neurostimulation devices will use a smartphone-based application (CAPTURE) to log real-world experiences while wearing additional sensors to record behavioral, physiological, and environmental data.

The study integrates multiple data modalities, including:

* Neural recordings from implanted neurostimulation devices
* Wearable sensor data, including:
* Audio-visual recordings
* GPS location tracking
* Accelerometry for movement analysis
* Autonomic physiology measurements (e.g., heart rate, skin conductance)
* Eye-tracking data

By synchronizing these data streams, researchers will establish a high-fidelity representation of autobiographical memory encoding and retrieval processes in daily life.

Analytic Methods and Data Integration

This study aims to develop computational frameworks for real-time data alignment and analysis. The primary methodological goals include:

* Temporal synchronization of multimodal data with neural recordings
* Automated feature extraction from behavioral and physiological data
* Neural signal processing techniques to identify patterns of activity associated with memory formation and retrieval
* Development of machine learning models to predict successful memory encoding and recall based on neural and behavioral signals
* These analytic advancements will enable researchers to assess memory-related brain activity in naturalistic environments, providing insights into the neural correlates of real-world autobiographical memory.

Potential Impact:

The findings from this study have significant implications for neuroscience, cognitive psychology, and clinical applications. By establishing methods for naturalistic neural recording and analysis, this research paves the way for neuromodulation-based memory enhancement therapies for individuals with memory disorders, including those with epilepsy, traumatic brain injury, and neurodegenerative diseases. The study also advances real-world cognitive neuroscience, enabling a deeper understanding of how the brain supports memory outside of laboratory settings.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* healthy to minor cognitive impairment

Exclusion Criteria:

* younger than 18 years of age
* more than minor cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Intracranial EEG power in Theta Band | 4 days
  iEEG power in the theta band between 4-8 Hz, will be assessed to identify the real-world experience features that contribute to changes in this important neural power band for memory encoding.
Intracranial EEG power in Gamma Band | 4 days
  iEEG power in the gamma band between 30-100 Hz, will be assessed to identify the real-world experience features that contribute to changes in this important neural power band for memory encoding.
Intracranial EEG normalized aperiodic exponent | 4 days
  This feature of intracranial EEG will be assessed as a broadband state-level change in brain activity during the participant's real-world experiences.

SECONDARY OUTCOMES:
Eye fixation duration to remembered experiences | 4 days
  Using eye-tracking, we will use the duration in time participants fixate on remembered experiences as a measure of visual attention.

OTHER OUTCOMES:
Questionnaire on Attitudes Regarding Neuroethics | Day 1
  This is a survey for people with responsive neurostimulation (RNS) devices. We ask some general demographic information. Then we will ask questions about how patients feel about the sharing of various types of personal data and how much they care about privacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Neurosciences Center, University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided